CLINICAL TRIAL: NCT05826951
Title: Social Effects of Alcohol
Acronym: SEA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IRB22-1696; 5R01DA002812-35 (NIH)
Record Dates: First submitted 2023-03-30; First posted 2023-04-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Alcohol-alcohol (Experimental): Both conversation partners receive alcohol
  Interventions: Drug: Alcohol
- placebo-placebo (Placebo Comparator): Both conversation partners receive placebo
  Interventions: Drug: Placebo
- alcohol-placebo (Experimental): participant receives alcohol and conversation partner receives placebo
  Interventions: Drug: Alcohol
- placebo-alcohol (Experimental): participant receives placebo and conversation partner receives alcohol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alcohol — Alcohol (0.8g/kg)
  Arms: Alcohol-alcohol; alcohol-placebo
Drug: Placebo — Placebo
  Arms: placebo-alcohol; placebo-placebo

SUMMARY:
In this study the investigator will assess the effect of a moderate dose of alcohol on emotional responses and feelings of connection during a dyadic semi-structured social interaction

DETAILED DESCRIPTION:
The study will use a within-subject crossover design with four sessions, in which participants receive alcohol or placebo across sessions. During the four sessions, the participants will engage in a conversation with a stranger, and emotional responses and feelings of connection will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* non-problem alcohol consumption of 2-20 drinks per week
* high school diploma or equivalent
* BMI between 19 and 26
* verbal fluency in English

Exclusion Criteria:

* High blood pressure
* Any medical condition requiring regular medication
* Individuals with a current (within the last year) DSM-IV Axis 1 diagnosis
* Women who are pregnant or trying to become pregnant.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
facial emotional responses | during the length of the conversation (45 min)
  alterations in the rate of positive facial expressions during the conversation, measured by muscle action units. These will be compared between the drug and placebo sessions
self-reported feelings of connection | at the end of each session (3.5 hrs post-drug administration). Changes across sessions will be assessed
  self-other overlap measure ratings 1-7, greater ratings indicates greater feelings of connection

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States